CLINICAL TRIAL: NCT04071431
Title: A Self-rating Risk Factor Questionnaire for the Improvement of Endoscopic Prediction of Gastrointestinal Cancer: a Big-data-based Diagnostic Study
Brief Title: A Questionnaire for Endoscopic Prediction Improvement of Gastrointestinal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yanqing Li (Other)
Responsible Party: Sponsor-Investigator, Yanqing Li, Professor, Shandong University
Organization: Shandong University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Screening
Other Study IDs: 2019SDU-QILU-08
Record Dates: First submitted 2019-08-24; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Early Detection of Cancer
Keywords: Early Detection of cancer; Gastrointestinal Neoplasms; Endoscopy, Gastrointestinal
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): During the application stage of endoscopy, the patients are required to complete a RFQ according to their own situations. The RFQs will soon uploaded to the core server of the quality control system and be analysed automatically immediately after finish. The results are sorted into four types including "N/A", "High-risk for esophageal cancer", "High-risk for gastric cancer" and "High-risk for colorectal cancer", which will be shown during the endoscopy of the specific person.
  The endoscopies are carried out by experienced endoscopists. All of the data of the endoscopy itself are collected and recorded in the quality control system.
  The RFQ results of this group are not known (deliberately showing "N/A") by the endoscopists before and during the endoscopy.
- Risk shown (Experimental): During the application stage of endoscopy, the patients are required to complete a RFQ according to their own situations. The RFQs will soon uploaded to the core server of the quality control system and be analysed automatically immediately after finish. The results are sorted into four types including "N/A", "High-risk for esophageal cancer", "High-risk for gastric cancer" and "High-risk for colorectal cancer", which will be shown during the endoscopy of the specific person.
  The endoscopies are carried out by experienced endoscopists. All of the data of the endoscopy itself are collected and recorded in the quality control system.
  The RFQ results of this group are known by the endoscopists before and during the endoscopy.
  Interventions: Other: Result masking

INTERVENTIONS:
Other: Result masking — The quality control system randomly shows the RFQ result to the endoscopists and keep 50% of the RFQ results are not known (deliberately showing "N/A") by the endoscopists before and during the endoscopy.
  Arms: Risk shown

SUMMARY:
Despite improvements in a range of chemo, radio and surgical therapies, the overall survival at 5 years from gastrointestinal cancer remains poor. Endoscopic early diagnosis is a key strategy to improve survival but the detection rate of early cancer varies among different countries. Risk factor questionnaire result is easy to be obtained and may be of great help for improving the detection rate. The aim of this research is to validate a risk factor questionnaire to help predict gastrointestinal cancer therefore allowing earlier diagnosis and higher detection rate.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged more than 18 years with or without GI symptoms attending for endoscopy.

Exclusion Criteria:

* Patients unable to cooperated the endoscopy or unable to complete it. People with endoscopy contraindications are naturally excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34906 (Estimated)
Dates: Start 2019-05-29 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Rate change | up to 24 months
  The endoscopic detection rate change of precancerous lesions and early GI cancer with the help of self-rating RFQ for the prediction of GI cancer.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China